CLINICAL TRIAL: NCT00850499
Title: A Randomized, Open-Label, Multicenter Phase 2 Study of VELCADE With Fludarabine in Comparison to Rituximab With Fludarabine in Follicular Lymphoma Patients Previously Treated With Rituximab
Brief Title: Phase 2 Study of VELCADE With Fludarabine in Comparison to Rituximab With Fludarabine in Follicular Lymphoma Patients Previously Treated With Rituximab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26866138-LYM-2033
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Results first posted 2012-11-01 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — fludarabine; Rituximab; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VELCADE and fludarabine (Group A) (Experimental): VELCADE 1.6 mg/m2 intravenously (IV) on Days 1, 8, 15, and 22 and fludarabine 40mg/m2/day orally on Days 1 to 5 of every 35-day cycle
  Interventions: Drug: fludarabine; Drug: VELCADE
- fludarabine and rituximab (Group B) (Active Comparator): fludarabine 40mg/m2/day orally on Days 1 to 5 and rituximab 375mg/m2 on Day 1 of every 35-day cycle
  Interventions: Drug: fludarabine; Drug: rituximab

INTERVENTIONS:
Drug: fludarabine — fludarabine 40mg/m2/day orally on Days 1 to 5 of every 35-day cycle
Drug: rituximab — rituximab 375mg/m2 on Day 1 of every 35-day cycle
  Arms: fludarabine and rituximab (Group B)
Drug: VELCADE — 1.6 mg/m2 intravenously (IV) on Days 1, 8, 15, and 22 of every 35-day cycle
  Arms: VELCADE and fludarabine (Group A)

SUMMARY:
This is a randomized, open-label, active-control, multicenter Phase 2 study of VELCADE+fludarabine in comparison with rituximab+fludarabine in subjects with relapsed advanced follicular lymphoma. Eligible subjects will be randomized in a 1:1 ratio between the 2 treatment arms (55 subjects per arm).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years or older
* Histologically proven diagnosis of follicular non-Hodgkin's lymphoma grades 1or 2 according to the World Health Organization classification
* Subjects must have received at least 12 doses (375mg/m2 or appropriately adjusted dose) of rituximab for the treatment of this lymphoma as single agent rituximab or in rituximab-containing regimens as documented in the subject's medical record
* Documented relapse or progression following last antineoplastic treatment
* At least 1 measurable tumor mass (≥1.5 cm x ≥1.0 cm)

Exclusion Criteria:

* Subjects with histological or clinical transformation to an aggressive lymphoma

  * prior treatment with VELCADE or fludarabine.
  * antineoplastic (including unconjugated therapeutic antibodies), experimental, or radiation therapy within 3 weeks before randomization
  * nitrosoureas within 6 weeks before randomization
  * radioimmunoconjugates or toxin immunoconjugates within 10 weeks before randomization
  * major surgery within 3 weeks before randomization
  * chronic use of corticosteroids, such as dexamethasone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (43):
- France (7):
  - CHU d'Amiens, Amiens
  - Institut Bergonie, Bordeaux
  - CHU Hotel Dieu, Clermont-Ferrand
  - Centre Victor Hugo, Le Mans
  - CHU Caremeau, Nîmes
  - Hoptial Saint Louis, Paris Cedex 10, 75
  - Hopital Cochin, Paris, 75, Cedex 14
- Germany (15):
  - Klinikum Bamberg, fachbereich 3, Bamberg
  - Charite, group Benjamin Franklin, Berlin
  - Hospital Spandau, Berlin
  - Vivantes Klinikum am Urban, Berlin, BE
  - Universitaetsklinikum Frankfurt, Frankfurt
  - Universitatsklinikum Gottingen, zentrum Innere medicin, Göttingen
  - Evangelisches Krankenhaus Hamm, Hamm
  - Klinikum Idar-Oberstein GmbH, Idar-Oberstein
  - Universitaetsklinikum Jena, Jena
  - Universitaetsklinikum Leipzig, Leipzig
  - Universitaetsklinikum Mainz, Mainz
  - Robert Bosch Krankenhaus, Stuttgart
  - Mutterhaus der Borromaeerinnen, Trier
  - Universitatsklinikum Ulm, Ulm
  - Klinikum der Stadt Villinger-Schwenningen, Villingen-Schwenningen
- Greece (2):
  - Laiko Hospital - 1st Dept. of Propaedeutic Internal Medicine, Athens
  - University Hospital of Heraklion- Department of Hematology, Heraklion- Crete
- Israel (5):
  - Haemek Medical Center - Hematology Department, Afula
  - Rambam Med.Center - Hematology Institute, Haifa
  - Hadassah University Hospital - Hematology Department, Jerusalem
  - Rabin Medical Center - Hematology Institute, Petah Tikva
  - Sheba MC - Hematology Institute, Ramat Gan
- Italy (10):
  - Policlinico di Bari, Bari
  - Istituto Di Ematologia E Oncologia Medica - L.A. Seragnoli - Policlinico S.Orsola Malpighi, Bologna
  - Clinica di Ematologia DIMI - A.O. Ospedale S. Martino, Genova
  - Ospedale Niguarda Ca' Granda, Milan
  - Azienda Ospedaliera Antonio Cardarelli, Napoli
  - Ospedale Policlinico San Matteo Irccs, Pavia
  - A.O.Univ.Pisana-Osp. Santa Chiara, Pisa
  - Università La Sapienza, Dipartimento di Biotecnologie Cellulari ed Ematologia, Via Benevento, 6, Roma
  - Azienda Ospedaliera Santa Maria di Terni, Terni
  - Divisione di Ematologia Ospedale San Bortolo - Hematology, Vicenza
- Spain (3):
  - Hospital Puerta del Mar, Secretaría de Hematología, 1ª planta, Cadiz
  - Hospital General Universitario Morales Meseguer, Secretaría de Hematología, 1ª planta, Murcia
  - Hospital Clinico Universitario Salamanca, Servicio de Hematología, 4º Planta, Salamanca
- Kantonsspital St.Gallen Department of Oncology/Hematology, Sankt Gallen, Switzerland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Velcade + Fludarabine | Rituximab + Fludarabine
Started | 4 | 8
Completed | 1 | 6
Not Completed | 3 | 2
Not completed — Adverse Event | 3 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Velcade + Fludarabine | Rituximab + Fludarabine | Total
Number analyzed (Participants) | 4 | 8 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 9
  >=65 years | 1 | 2 | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 61.3 (12.84) | 60.0 (10.06) | 60.4 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  France | 0 | 3 | 3
  Greece | 0 | 1 | 1
  Spain | 1 | 0 | 1
  Israel | 1 | 0 | 1
  Germany | 0 | 1 | 1
  Switzerland | 1 | 0 | 1
  Italy | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: The proportion of response-evaluable subjects who achieved a confirmed complete response (CR) or complete response unconfirmed (CRu). Disease response and progression were evaluated according to modified International Workshop Response Criteria (IWRC) criteria by radiographic imaging and other procedures as necessary.
Time Frame: Up to 8 cycles (1 cycle is 35 days: 280 days)
Population: Received at least one dose of study drug
Measure: Number; unit: participants
Groups:
- Velcade + Fludarabine: Velcade + Fludarabine
- Rituximab + Fludarabine: Rituximab + Fludarabine
Arm/Group | Velcade + Fludarabine | Rituximab + Fludarabine
Number analyzed (Participants) | 4 | 8
participants | 2 | 3

2. Secondary Outcome: Overall Response Rate
Description: The proportion of subjects who achieve CR, CRu, or partial response (PR) relative to the response evaluable population. Disease response and progression were evaluated according to the modified IWRC criteria by radiographic imaging and other procedures as necessary.
Time Frame: Up to 8 cycles (1 cycle is 35 days: 280 days)
Population: Received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | Velcade + Fludarabine | Rituximab + Fludarabine
Number analyzed (Participants) | 4 | 8
participants | 3 | 6

ADVERSE EVENTS:
Arm/Group | Velcade + Fludarabine | Rituximab + Fludarabine
Serious Adverse Events (participants affected / at risk) | 2/4 | 2/8
Other Adverse Events (participants affected / at risk) | 4/4 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Velcade + Fludarabine (N=4) | Rituximab + Fludarabine (N=8)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Dypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Respiratory gas exchange disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Velcade + Fludarabine (N=4) | Rituximab + Fludarabine (N=8)
Leukopenia (Blood and lymphatic system disorders) | 1 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3
Blepharitis (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 1 | 3
Fatigue (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 0 | 1
Performance status decreased (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Tinea infection (Infections and infestations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Conversion disorder (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No